CLINICAL TRIAL: NCT02968797
Title: SafeSed Validation Study, Comparing Performance to Capnography, as a Monitoring Technology of Respiratory Parameters
Brief Title: Clinical Comparative Study to Validate Performance of SafeSed Prototype Monitoring Endoscopy Under Sedation
Acronym: SafeSed
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0143-16-MMC
Record Dates: First submitted 2016-09-07; First posted 2016-11-21 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SafeSed — Monitor respiratory parameters

SUMMARY:
SafeSed prototype monitors respiratory parameters by tracking chest movements with optical and accelerometer markers. The respiratory parameters are compared to respiratory parameters measured by a spirometer and a capnograph.

DETAILED DESCRIPTION:
Patients performing endoscopy procedures under sedation at the gastro clinic will be monitored by SafeSed in addition to being monitored by capnography, used by an anaesthetist. All patients will be monitored using the same two techniques (SafeSed and Capnography). No clinical decisions will be made based upon the data generated by the SafeSed system.

The data from all sources will be compared (post factum) to validate SafeSed performance.

The data collected on the SafeSed prototype will not be used for treatment of the patient.

The comparative analysis will be free vto be used by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* class 1-3 per American Society Anesthesiologists Physical Status Classification
* Subject signed Informed Concent Form

Exclusion Criteria:

* Pregnancy
* Unresolved pulmonary infection requiring active treatment
* Chronic pulmonary disease
* Any othe medical condition, that treating physician determines participating in the study is unadvisable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to perform endoscopy procedures under sedation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparative data of monitoring respiratory by 2 technologies | 4 months
  Validation of SafeSed performance by comparing to capnography. The respiratory rate (RR) and end tidal carbon dioxide (ETCO2) levels will be collected into a personal computer, and stored with a continuous time-stamp. RR, tidal volume (TD) and minute ventilatio (MV) calculations using the SafeSed markers chest movements will be stored at the same PC using the same time-stamp. Comparison will show correlation between deterioration events of respiratory parameters. This comparison will be the outcome of off-line analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Fredman, MD, Principal Investigator — Israel: Clalit Health bServices
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No